CLINICAL TRIAL: NCT04899596
Title: High Risk Factor, Clinical Feature, and Follow up of Neonatal Arrhythmia
Status: Completed | Type: Observational
Sponsor: Daping Hospital and the Research Institute of Surgery of the Third Military Medical University (Other)
Collaborators: Children's Hospital of Chongqing Medical University (Other)
Responsible Party: Principal Investigator, Chen Long,MD, Daping Hospital and the Research Institute of Surgery of the Third Military Medical University, Daping Hospital and the Research Institute of Surgery of the Third Military Medical University
Other Study IDs: arrhythmia
Record Dates: First submitted 2021-05-05; First posted 2021-05-24 (Actual); Last update posted 2021-05-24 (Actual); Status verified 2021-05

CONDITIONS: Neonatal Arrhythmia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
This study included 189 newborns (77 male,112 female) diagnosed with arrhythmia in the NICU of Children's Hospital of Chongqing Medical University, China, from January 2015 through December 2019. To investigate the high-risk factors, clinical manifestations, and clinical outcomes of neonatal arrhythmia.

DETAILED DESCRIPTION:
The incidence of neonatal arrhythmia is 3.94‰(189/47911), and the mortality of neonatal arrhythmia is 0.21‰(10/47911) within 1 year after birth.

ELIGIBILITY:
Inclusion Criteria:①Newborns admitted in the Department of Neonatology of Children's Hospital Affiliated to Chongqing Medical University from January 2015 to December 2019;② 12-lead ECG and/or 24-hour dynamic ECG suggest arrhythmias, including children with sinus tachycardia and sinus arrhythmia.

Exclusion Criteria:not have

Ages: 1 Minute to 28 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: neonates
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Electrocardiogram | up to 12 weeks
  A 12-lead electrocardiogram or dynamic electrocardiogram
anti-arrhythmia | before 1 year old
  Use antiarrhythmic medications
death | up to 12 weeks
  neonates died
death | before 1 year old
  neonates died
recurrence | before 1 year old
  Arrhythmia occurs again

CONTACTS AND LOCATIONS:
Locations (1):
- Daping Hospital and the Research Institute of Surgery of the Third Military Medical University, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided